CLINICAL TRIAL: NCT02776358
Title: High Fidelity Simulation (HFS) Versus Video-case(VC) Trainings in the Assessement and Management of Severe Asthma Attack Among Medical School Students: a Randomized Controlled Study
Brief Title: HFS in the Assessement and Management of Severe Asthma Attack Among Fifth Year Medical School Students
Acronym: SimAG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Clinical Professor, University of Monastir
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SimAG
Record Dates: First submitted 2016-05-04; First posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Fidelity Simulation (Experimental): Students will receive a 1 hour High fidelity simulation session
  Interventions: Other: High Fidelity Simulation
- Video Case (Experimental): Students will receive a 1 hour assisted Video Case learning session
  Interventions: Other: Video case

INTERVENTIONS:
Other: High Fidelity Simulation — A HFS session for an asthma attack require:
  * a 5 minutes briefing session: case and equipments presentation and choice of participants
  * 15 minutes of actual simulation
  * 40 minutes of debriefing
  A pre and a post test will be taken by the students before and after the session and a satisfaction questionnaire at the end of the course.
  Also, another test will be done after 7 days of the course.
  Arms: High Fidelity Simulation
Other: Video case — a video case (or video box) session in which students will attend a video-projection of a real case of an asthma attack and discuss with the trainer the different steps of the assessement and management of an asthma attack.
  A pre and a post test will be taken by the students before and after the session and a satisfaction questionnaire at the end of the course.
  Also, another test will be done after 7 days of the course.
  Arms: Video Case

SUMMARY:
Bedside clinical case learning, such for respiratory distress, represent a challenge for medical teachers, especially in critical conditions. In fact, this kind of learning implicate the presence of an appropriate case (the patient itself), framework and may be time consuming which could compromise the patient's safety and wellbeing.

New pedagogic tools have emerged to strengthen the medical reasoning and the acquisition of knowledge. in recent years, the development of medical simulation has found a growing interest in the medical teaching field. Contextualization, reproducibility and reliability are the characteristics of high-fidelity simulation (HFS) which guarantee a lifetime experience of clinical conditions without putting at risk patient's safety and comfort.

The aim of this study is to assess the impact of HFS on fifth year medical students learning skills in the assessement and management of an acute asthma attack in the emergency room, and to compares it to other modern teaching tools such as "video-case"

ELIGIBILITY:
Inclusion Criteria:

* all fifth year medical students allocated to the one month internship period in the emergency departement.

Exclusion Criteria:

* students refusing to participate in the protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Difference between the pre and the post-test scores in each group (delta Score) | Just before the teaching course (baseline) and one hour later
  The difference between the pre and the post-test scores is calculated as follow:
  delta score = post-test score - pre-test score

SECONDARY OUTCOMES:
Late performance score | 7 days after the teaching course
  This score is calculated based on a test taken 7 days after the teaching course to assess the students memory of the clinical case and acquired knowledge.
Level of satisfaction | one hour after the teaching course
  A five point likert scale is given to each student to assess their level of satisfaction regarding the teaching technique.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed habib Grissa, MD, Principal Investigator — Emergency Department , university hospital of Monastir, TUNISIA; Nouira Semir, Professor, Principal Investigator — Emergency Department , university hospital of Monastir, TUNISIA
Locations (1):
- university of Monastir, Monastir, Monastir Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grissa MH, Dhaoui R, Bel Haj Ali K, Sekma A, Toumia M, Sassi S, Sakly AK, Zorgati A, Bouraoui H, Ben Soltane H, Mezgar Z, Boukef R, Boubaker H, Bouida W, Beltaief K, Nouira S. Comparison of simulation and video-based training for acute asthma. BMC Med Educ. 2023 Nov 16;23(1):873. doi: 10.1186/s12909-023-04836-7. PMID 37974223